CLINICAL TRIAL: NCT00545623
Title: Acupuncture and Relaxation Response for GI Symptoms and HIV Medication Adherence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Bei-Hung Chang, Associate Professor, Boston University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT003377-01 (NIH); R21AT003377-01 (NIH)
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; Alternative Medicine; Complementary Medicine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ACU+RR (Active Comparator): acupuncture + relaxation response CD
  Interventions: Procedure: Acupuncture; Behavioral: Relaxation Response
- SHAM+RR (Active Comparator): sham acupuncture + relaxation response CD
  Interventions: Behavioral: Relaxation Response
- ACU+EDU (Active Comparator): acupuncture+control CD
  Interventions: Procedure: Acupuncture
- SHAM+EDU (Sham Comparator): sham acupuncture+control CD
  Interventions: Other: sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — acupuncture twice/week for the first 4 weeks and once/week for another 4 weeks
  Arms: ACU+EDU; ACU+RR
Behavioral: Relaxation Response — listening to CDs with verbal instructions of techniques to elicit relaxation response
  Arms: ACU+RR; SHAM+RR
Other: sham acupuncture — sham acupuncture twice/week for the first 4 weeks and once/week for another 4 weeks
  Arms: SHAM+EDU

SUMMARY:
The aims of the study are to investigate individual, combined and added effects of acupuncture and the relaxation response in reducing gastrointestinal symptoms, improving medication adherence and quality of life among people living with HIV/AIDS. The study will also explore the mechanism of these therapeutic effects of acupuncture and the relaxation response.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV-positive status or AIDS diagnosis
2. Self report of having at least one of the 6 GI symptoms: diarrhea, loose stools, gas/flatulence or bloating, abdominal pain, nausea, or vomiting that have persisted for at least 8 weeks.
3. Being on a stable antiretroviral regimen containing Nucleoside/nucleotide reverse transcriptase inhibitors and/or protease inhibitors- for at least 8 weeks.

Exclusion Criteria:

1. Incident diagnosis of any of the following conditions within the past month or during study period: Pneumocystis carinii pneumonia, Kaposi's sarcoma, Mycobacterium avian complex, Cytomegalovirus, Non-Hodgkins lymphoma, Lymphoma or other cancer, Pelvic inflammatory disease, AIDS-related dementia, Bacterial or other infection, Diabetes, Acute moderate or severe neutropenia, Cryptococcus, Progressive multifocal leukoencephalopathy, Idiopathic thrombocytopenic purpura. All of these conditions are major opportunistic infections or medical complications that may require hospitalization and additional pharmaceutical intervention.
2. GI diagnoses of irritable bowel syndrome, Crohn's Disease, parasites, any type of gastric ulcer or ulcerative colitis or cancer in any part of the gastrointestinal system. These are conditions not related to HIV diagnosis and could result in digestive problems similar to those we are investigating.
3. Onset of acute opportunistic infection.
4. Hemophilia or other bleeding disorder since that will make acupuncture treatment unsafe.
5. Pregnant women will be excluded since, although none of the acupuncture points or combinations are contraindicated in pregnancy, the presence of morning sickness could serve as a potential confounding factor.
6. Current users of acupuncture for treating GI symptoms.
7. Current practice of relaxation response.
8. Current enrollment in another clinical intervention study.
9. Cognitive impairment as measured by Mini Mental Status Examination (MMSE), a reliable and valid screening instrument for the detection of cognitive impairment, using a commonly used cut-off point of 24.
10. If use of Chinese herbs has been recently discontinued, a potential participant must have at least 2 weeks without herb use to be eligible for the study. Because use of herbs is occasionally accompanied by digestive disorders,a period of stabilizing is required before acupuncture treatment can be initiated. This washout period has been conservatively estimated by ACP staff herbalists to constitute a sufficient time for effects of herbs to cease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bei-Hung Chang, Sc.D., Principal Investigator — Boston University
Locations (1):
- Pathways to Wellness, Boston, Massachusetts, United States

REFERENCES:
- [Result] Chang BH, Sommers E. Acupuncture and the relaxation response for treating gastrointestinal symptoms in HIV patients on highly active antiretroviral therapy. Acupunct Med. 2011 Sep;29(3):180-7. doi: 10.1136/acupmed-2011-010026. Epub 2011 Jun 24. PMID 21705396

RESULTS

PARTICIPANT FLOW:
Groups:
- ACUP+RR: acupuncture + relaxation response CD
  Acupuncture: acupuncture twice/week for the first 4 weeks and once/week for another 4 weeks
  Relaxation Response: listening to CDs with verbal instructions of techniques to elicit relaxation response
- ACUP+EDU: acupuncture+education CD
  Acupuncture: acupuncture twice/week for the first 4 weeks and once/week for another 4 weeks
- SHAM+EDU: sham acupuncture+education CD
  sham acupuncture: sham acupuncture twice/week for the first 4 weeks and once/week for another 4 weeks
Period: Overall Study
Arm/Group | ACUP+RR | SHAM+RR | ACUP+EDU | SHAM+EDU
Started | 32 | 31 | 33 | 34
Completed | 25 | 21 | 20 | 23
Not Completed | 7 | 10 | 13 | 11

BASELINE CHARACTERISTICS:
Population: A total of 15 patients did not start the intervention after enrollment, 1, 4, 6, and 4 patients in ACUP+RR, SHAM+RR, ACUP+EDU, and SHAM+EDU arms respectively. As such there are a total of 115 patients with baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACUP+RR | SHAM+RR | ACUP+EDU | SHAM+EDU | Total
Number analyzed (Participants) | 31 | 27 | 27 | 30 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (8.8) | 45.0 (7.1) | 47.1 (9.9) | 47.0 (8.2) | 46.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 7 | 9 | 34
  Male | 22 | 18 | 20 | 21 | 81
Region of Enrollment [Number; unit: participants]
  United States | 31 | 27 | 27 | 30 | 115

OUTCOME MEASURES:

1. Primary Outcome: Changes in GI Symptom Per Intervention Session
Description: We used the GI symptom subscale of the Revised HIV Sign and Symptom Checklist (SSC-HIV) to measure the intensity (0-10) of the six targeted GI symptoms: diarrhea, loose stools, gas/bloating, abdominal pain, nausea and vomiting, with 0 indicating no symptom and 10 indicating most sever symptom. Rating changes per intervention session were estimated using a mixed effects regression model controlling for baseline ratings. Data of loose stools are presented here.
Time Frame: 8 weeks
Population: An intent-to-treat approach was used for analysis. That is all patients who had at least one data points were included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACUP+RR | SHAM+RR | ACUP+EDU | SHAM+EDU
Number analyzed (Participants) | 27 | 25 | 25 | 27
units on a scale | -0.24 (0.04) | -0.08 (0.04) | -0.09 (0.04) | -0.09 (0.04)

ADVERSE EVENTS:
Time Frame: 8 week study intervention period and 6 month follow up period
Arm/Group | ACUP+RR | SHAM+RR | ACUP+EDU | SHAM+EDU
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 5/32 | 5/31 | 5/33 | 2/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACUP+RR (N=32) | SHAM+RR (N=31) | ACUP+EDU (N=33) | SHAM+EDU (N=34)
pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
broken hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
thrush (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
car accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abnormal but benign tissue in descending colon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sever esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
kidney problem (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
basal cell CA surgery (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
stomach virus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No